CLINICAL TRIAL: NCT04461132
Title: Investigation of the Effect of Manual Lymphatic Drainag on Venous Ulcer Healing Rate
Brief Title: The Effect of Manual Lymphatic Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Collaborators: Istanbul Health Sciences University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2017.209
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Venous Leg Ulcer; Venous Insufficiency; Lymphatic Disease
MeSH Terms: conditions — Varicose Ulcer; Venous Insufficiency; Lymphatic Diseases | interventions — Manual Lymphatic Drainage; Skin Care; Exercise

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Lymphatic Drainage Group (Active Comparator): All patients were treated 3 times a week for 4 weeks. The treatment program of these patients included manual lymphatic drainage on the leg, skin care, bandaging and exercise.
  Interventions: Other: Manual Lymphatic drainage (MLD); Other: Skin Care; Other: Exercise
- Shame Manual Lymphatic Drainage Group (Sham Comparator): All patients were treated 3 times a week for 4 weeks. The treatment program of these patients included shame manual lymphatic drainage on the leg, skin care, bandaging and exercise. Shame manual lymphatic drainage include light touches instead of real manual lymphatic drainage techniques
  Interventions: Other: Skin Care; Other: Exercise; Other: Shame Manual Lymphatic drainage

INTERVENTIONS:
Other: Manual Lymphatic drainage (MLD) — MLD vith vodder technique was applied to leg
  Arms: Manual Lymphatic Drainage Group
Other: Skin Care — Wound was cleaned with salin and covered by dressing without including active products
Other: Exercise — breathing and foot pump exercise was prescribed
Other: Shame Manual Lymphatic drainage — manual lymphatic drainage was applied with light touch instead of real mld techniques
  Arms: Shame Manual Lymphatic Drainage Group

SUMMARY:
In venous ulcer, venous insufficiency is accompanied by lymphatic insufficiency. Manual lymphatic drainage (mld) technique cause to increase contraction rate of lymphatic collector and venous flow. It is known that Manual lymphatic drainage accelerates microcirculation, enabling nutrients and oxygen to reach tissues and at the same time removing residual substances from the tissue. We hypothesis that if we inrease to lypmhatic activity with MLD, we could stimulate healing of ulcer. The aim of this study to investigate the effect of manual lymphatic drainage on venous ulcer healing.

ELIGIBILITY:
Inclusion Criteria:

* with venous ulcer unhealing for at least 6 weeks
* Without enfection
* vascular surgery is not indicated
* There is no obstruction to apply MLD and compression to lower extremty

Exclusion Criteria:

* with diabetic mellutus
* with enfection
* with ABI<0,7
* Patients who have undergone venous vascular surgery
* Patients undergoing active wound closure treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of wound healing | Change from baseline wound healing following the end of treatment (12. treatment session) and 1 month after the end of treatment.
  Wound was assesed by analyzing photographes of wound with Tracker software.
Evaluation of range of motion of ankle | Change from baseline range of motion following the end of treatment (12. treatment session) and 1 month after the end of treatment.
  range of motion of ankle was measured with goniometer
Evaluation of pain | Change from baseline pain following the end of treatment (12. treatment session) and 1 month after the end of treatment.
  Pain was evaluated by Visual Analog Scale between 0 (no pain)-10 (extreme) pain.
evaluation of edema | Change from baseline edema following the end of treatment (12. treatment session) and 1 month after the end of treatment.
  edema was measured by 3D scanner
evaluation of quality of life | Change from baseline quality of life following scores the end of treatment (12. treatment session) and 1 month after the end of treatment.
  quality of life was evaluated by SF- 12

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Kablan, PhD, Study Director — University of Health science
Locations (1):
- Istanbul Saglık Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Azoubel R, Torres Gde V, da Silva LW, Gomes FV, dos Reis LA. [Effects of the decongestive physiotherapy in the healing of venous ulcers]. Rev Esc Enferm USP. 2010 Dec;44(4):1085-92. doi: 10.1590/s0080-62342010000400033. Portuguese. PMID 21337794
- [Result] Crawford JM, Lal BK, Duran WN, Pappas PJ. Pathophysiology of venous ulceration. J Vasc Surg Venous Lymphat Disord. 2017 Jul;5(4):596-605. doi: 10.1016/j.jvsv.2017.03.015. PMID 28624002
- [Result] de Roos KP, Wittens CH, Maessen-Visch MB, van der Wegen-Franken CP. [Universal Dutch guideline on 'Venous disease']. Ned Tijdschr Geneeskd. 2014;158(0):A8076. Dutch. PMID 27707417
- [Result] Williams A. Manual lymphatic drainage: exploring the history and evidence base. Br J Community Nurs. 2010 Apr;15(4):S18-24. doi: 10.12968/bjcn.2010.15.Sup3.47365. PMID 20559172
- [Result] Kelechi TJ, Johnson JJ, Yates S. Chronic venous disease and venous leg ulcers: An evidence-based update. J Vasc Nurs. 2015 Jun;33(2):36-46. doi: 10.1016/j.jvn.2015.01.003. PMID 26025146
- [Result] Hampton S. An introduction to various types of leg ulcers and their management. Br J Nurs. 2006 Jun 8-21;15(11):S9-13. doi: 10.12968/bjon.2006.15.Sup2.21235. PMID 16835515